CLINICAL TRIAL: NCT06745297
Title: A Two-part, Randomised, Single-blind, Placebo-controlled, Single and Multiple Rising Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of BI 3776528, Administered to Healthy Male Participants
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 3776528 Are Tolerated
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1526-0001; 2024-515222-92-00 (EU CTIS Number); U1111-1307-8288 (Other: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-12-19; First posted 2024-12-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This trial will be conducted in 2 parts: Part 1 (single doses) and Part 2 (multiple doses). Part 1 comprises of 2 subparts: Parts 1a and 1b.
  Part 1b starts only after the dose has been tested in part 1a and was safe and of acceptable tolerability.
  Part 2 of the study will only commence after the successful administration of the planned dose to the last subject in part 1a.
Who Masked: Participant
Masking Description: Part 1a of this trial is a randomized, single-blind, and placebo-controlled. Part 1b of the trial is randomized, open-label, and with a two-way crossover design.
  Part 2 of the trial is single-blind, randomized, and placebo-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: BI 3776528; Drug: short-acting benzodiazepine
- Placebo group (Placebo Comparator): Applicable for part 1a and part 2 of the trial.
  Interventions: Drug: Placebo matching BI 3776528; Drug: short-acting benzodiazepine

INTERVENTIONS:
Drug: BI 3776528 — BI 3776528
  Arms: Treatment group
Drug: Placebo matching BI 3776528 — Placebo matching BI 3776528
  Arms: Placebo group
Drug: short-acting benzodiazepine — short-acting benzodiazepine

SUMMARY:
The trial aims to study the safety, tolerability, and pharmacokinetics of single and multiple rising doses of BI 3776528.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination and clinical laboratory.
2. Age of 18 to 50 years (inclusive)
3. BMI of 18.5 to 29.9 kg/m² (inclusive), body weight above 60 kg (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Exclusion criteria:

1. Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement at screening of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the (age-adapted) reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin), renal parameters (creatinine) exceeding the upper limit of normal (ULN) after repeated measurements or abnormal thyroid stimulating hormone (TSH) values outside of the normal range after repeated measurements.
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Part 1a and Part 2: Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 62 days
Part 1b: AUC0-tz of BI 3776528 in plasma (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 27 days
Part 1b: Cmax of BI 3776528 in plasma (maximum measured concentration of the analyte in plasma) | up to 27 days

SECONDARY OUTCOMES:
Part 1a: AUC0-∞ of BI 3776528 in plasma (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 27 days
Part 1a: Cmax of BI 3776528 in plasma | up to 27 days
Part 1b: AUC0-∞ of BI 3776528 in plasma | up to 27 days
Part 2: AUCτ,ss of BI 3776528 in plasma (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 27 days
Part 2: Cmin,ss of BI 3776528 in plasma (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 27 days
Part 2: Cmax,ss of BI 3776528 in plasma (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 27 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com